CLINICAL TRIAL: NCT06080685
Title: Efficacy of Character Strengths Intervention in Enhancing Character Strengths and Self-esteem Among Adolescents
Acronym: (CSI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Asma Rashid, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: FJWU/EC/2023/61; FJWU/EC/2023/61 (Other: FJWU)
Record Dates: First submitted 2023-09-27; First posted 2023-10-12 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Mental Health Issue; Mutism; Orthopedic Disorder
Keywords: Adolescents with physical disability
MeSH Terms: conditions — Mutism; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Who receives intervention. Character strengths intervention will be administered in 5 sessions.
  Interventions: Behavioral: Character Strengths Intervention
- Waitlist Control Group (Active Comparator): Who would receive the intervention after the study completion.
  Interventions: Behavioral: Character Strengths Intervention

INTERVENTIONS:
Behavioral: Character Strengths Intervention — Session 1. Getting Started: Introducing and Exploring Character Strengths Session 2. Boost a Lower Strength Session 3. Cultivate your inner self + Loving-Kindness Meditation Session 4. Gratitude Letter + Three Good things Session 5. Conclusion Each session will consist of 1-hour, which will be delivered once a week for 5 weeks. Moreover, participants will be given homework which they will practice the rest of the week.
  Other Names: Positive Psychology Interventions

SUMMARY:
The goal of this study is to better understand the experiences of adolescents with physical disabilities and assess the effectiveness of a Character Strengths Intervention (CSI) in improving their self-esteem, character strengths, and mental health. We will also compare these outcomes between two groups: one receiving the intervention and the other not receiving any treatment.

Main Research Questions:

How do adolescents with physical disabilities perceive their self-esteem, character strengths, and mental health, including psychological adjustment, psychological distress, psychological wellbeing, life satisfaction, and resilience? Can the Character Strengths Intervention (CSI) enhance the self-esteem, character strengths, and mental health (psychological adjustment and distress) of adolescents with physical disabilities?

Study Tasks:

Participants, who are adolescents aged 12-18 years, will be asked to provide informed consent to participate in the study.

They will complete questionnaires to assess their self-esteem, character strengths, and mental health as a pre-assessment.

Participants in the intervention group will undergo the Character Strengths Intervention (CSI), which includes activities like exploring character strengths, writing gratitude letters, and practicing fresh look meditation, among others.

After the intervention, participants will complete post-assessment questionnaires to measure changes in self-esteem, character strengths, and mental health.

There will be a control group that does not receive any treatment.

Comparison Group:

Researchers will compare the outcomes between the intervention group, who received the Character Strengths Intervention (CSI), and the control group, who did not receive any treatment. This will help us determine if the intervention had a significant impact on self-esteem, character strengths, and mental health outcomes for adolescents with physical disabilities.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents with physical disability
2. Adolescents with physical disability in the age range 11-18
3. Rural and urban residences
4. Urdu, Englishspeaking
5. Rawalpindi and Islamabad special education schools

Exclusion Criteria:

1. Adolescents under age 11 and above 18
2. Adolescents whose parents, teachers, or themselves would not be agreed and signed informed consent to participate in the study would be excluded
3. Adolescents with physical disability such as:

   * Sensory disability (mute and Fully/partial-visual impairment) impairment
   * Hearing impairment
   * Deaf-blindness
   * And intellectual and cognitive impairment
4. Adolescents with severe psychiatric and major medical issues -

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2023-09-23 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Self-esteem | 1 month
  10-item scale "Rosenberg Self-esteem Scale" used to measure.
Character strengths | 1 month
  98 items scale "The Values in Action (VIA) Youth Survey" is used.

SECONDARY OUTCOMES:
Psychological wellbeing | 1 month
  14 Items scale "the Warwick-Edinburgh Mental Well-being Scale (WEMWBS)" is used to measure psychological wellbeing.
Life Satisfaction | 1 month
  5 items scale "Satisfaction with Life Scale" is used.
Resilience | 1 month
  10 items "Connor-Davidson Resilience Scale (CD-RISC-10)" is used.

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Directorate General of Specials Education, Islamabad, Captial
  - Al-Ghazali Special Education School, Rawalpindi, Punjab Province
  - Army Public Special Education Centre, Rawalpindi, Punjab Province